CLINICAL TRIAL: NCT06198881
Title: Association Between Labor Induction and Birth Weight in Cases of Fetal Macrosomia: The MACROMODA Cohort Study
Acronym: MACROMODA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5317
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Birth Weight; Macrosomia, Fetal
Keywords: macrosomia; labor induction; perineal tears; hemorrhage; full-term deliveries; singleton
MeSH Terms: conditions — Birth Weight; Fetal Macrosomia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- induction of labor: Patient having been induced by cervical ripening (prostin gel (2mg/24h), intravaginal prostaglandin (10mg/24h), balloon (<12h exposure time) or oral misoprostole (50µg/4h until induction of labor) or induction of contractions by oxytocin (gradual increase in dose) for suspected ultrasound macrosomia (according to the criteria of the DAME study)
- natural labor: Patient presenting with spontaneous labor after 37 weeks of gestation.

SUMMARY:
The rising prevalence fof fetal macrosomia represents a significant challenge in obstetrics, affecting both maternal and neonatal outcomes. Such challenges include complications like perineal tears and postpartum hemorrhage. Concurrently, the frequency of labor induction practices on the rise, yet the implications for neonatal weight are inadequately understood. To address this gap, our study aims to evaluate the association between labor induction and neontal birth weight through a population-based cohort study. The findings have the potential to inform more accurate clinical guidelines, thereby enhancing the quality of maternity care.

ELIGIBILITY:
Inclusion Criteria:

* Full-term deliveries (≥ 37 weeks of gestation)
* Singleton
* Birth weight > 4000g
* Complete medical records available for analysis

Exclusion Criteria:

* Delivery < 37 weeks
* Uterus > bi-scarred
* Presentation of the headquarters
* Maternal or fetal pathology modifying the route/time of delivery (pre-eclampsia, fetal heart rate abnormalities, cholestasis, chorioamnionitis, metrorrhagia, covering placenta, etc.)

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The selected patients are thoses who gave birth at term (>37 weeks) of a macrosome fetus (>4000g) in one of the maternity wards of the civil hospices of Lyon (Hospital de la Croix Rousse, Hopital Femme Mere Enfant or Hopital Lyon Sud). Patients are subsequently categorized based on whether their labor was induced or not. The characteristics of the pregnancy, the route of delivery and the fetal outcome are then collected in the computerized medical records and analyzed.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of vaginal deliveries among the population studied | during Delivery
  Number of vaginal deliveries among the population studied

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Femme-Mère-Enfant, Bron
  - Croix Rousse Hospital, Lyon
  - Hôpital Lyon Sud, Pierre-Bénite